CLINICAL TRIAL: NCT05947435
Title: The Effect of Use of Tranexamic Acid in Percutaneous Nephrolithotomy on Blood Loss and Surgical Visual Clarity
Brief Title: Tranexamic Acid in Percutaneous Nephrolithotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Berna Caliskan, M.D., Haseki Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 108-2021
Record Dates: First submitted 2023-07-07; First posted 2023-07-17 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Percutaneous Nephrolithotomy; Intraoperative Use of Tranexamic Acid
Keywords: blood loss; percutaneous nephrolithotomy; tranexamic acid; visual image quality
MeSH Terms: conditions — Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Randomisation was designed as 3 (n= 25) named Groups A, B, and Group C in a 1:1:1 ratio with a computer-based algorithm and sealed in opaque envelopes by the surgeon assigned to the study. The investigative anesthesiologist selected an envelope in the order of numbers on it, and Group A continued with an IV infusion of 10 mg/kg tranexamic acid for 20 minutes just before the surgical incision. In Group B, 10 mg/kg tranexamic acid was placed in the first irrigation solution, and in Group C, no drug was given in either way. The urologist was blind to the study groups and was the evaluator of an intraoperative visual score. Postoperative Hb and Hct values and complications were followed by the surgeons who were also blinded to the groups, and the decision of blood replacement was made according to the Hct values according to our standard protocol of the urology department.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tranexamic acid IV (Experimental): Group A received an IV infusion of 10 mg/kg tranexamic acid for 20 minutes just before the surgical incision.
  Interventions: Drug: Tranexamic acid
- Tranexamic acid irrigation (Experimental): 10 mg/kg tranexamic acid was placed in the first irrigation solution
  Interventions: Drug: Tranexamic acid
- Control (No Intervention): The control group did not receive tranexamic acid in either way

INTERVENTIONS:
Drug: Tranexamic acid — Tranexamic acid was administered in intravenous or locally within irrigation fluid
  Other Names: Transamin®
  Arms: Tranexamic acid IV; Tranexamic acid irrigation

SUMMARY:
Tranexamic acid, once a randomly used antifibrinolytic agent, has been in standard protocols for many specific surgeries. Studies are still needed to standardize the dose and route of tranexamic acid administration, examine its possible contributions in urological surgery, and establish a protocol for its use.

To contribute to this goal, the study was designed as a prospective, randomized, double-blind study on 75 patients with one control and 2 study groups (n=25) who underwent percutaneous nephrolithotomy. Group Tranexamic acid received 10 mg/kg intravenous tranexamic acid preoperatively. And Group Irrigation received the same amount in the initial irrigation fluid. Primarily,the total amount of blood transfusion and the changes in haemoglobin and haematocrit values during two postoperative days were observed. Distinctively, continuous intraoperative haemoglobin saturation was monitored. Secondarily, surgical visual clarity with a standard visual score was questioned to reveal its contribution to surgical practicality, operative time, and residual fragment quantity.

DETAILED DESCRIPTION:
The study was designed as a double-blind, prospective, randomised, controlled study after approval of our Institutional ethics committee (dossier no: 108-2021) and assessed patients scheduled for PCNL after January 2022 for eligibility. After obtaining written informed consent, 75 patients (3 groups; 1:1:1 distribution; n=25) were allocated, and the study was conducted in Haseki Training and Research Hospital until May 2023, with the principles outlined in the Helsinki Declaration.

Study subjects The study population was 18-70 years old and ASA I-III patients scheduled for PCNL surgery. Exclusion criteria were tranexamic acid hypersensitivity, history of subarachnoid haemorrhage, previous cerebrovascular event, a history of arterial-venous embolism or a tendency to thromboembolism, abnormal liver function tests, unstable cardiovascular disease, acute or chronic renal failure, presence of any haematological disease and known colour blindness.

Patient randomization and blindness Randomization was designed as 3 (n= 25) named Groups A, B, and Group C in a 1:1:1 ratio with a computer-based algorithm and sealed in opaque envelopes by the surgeon assigned to the study. The investigative anesthesiologist selected an envelope in the order of numbers on it, and Group A continued with an IV infusion of 10 mg/kg tranexamic acid for 20 minutes just before the surgical incision. In Group B, 10 mg/kg tranexamic acid was placed in the first irrigation solution; in Group C, no drug was given either way. The urologist was blind to the study groups and was the evaluator of an intraoperative visual score. Postoperative Hb and Hct values and complications were followed by the surgeons who were also blinded to the groups, and the decision of blood replacement was made according to the Hct values according to our standard protocol of the urology department.

Anaesthesia and surgical technique All surgeries were performed under general anaesthesia with standard monitorisation and non-invasive MASIMO Hemoglobin (SpHb®) real-time monitoring. After the ureteral catheter was placed, the patient was placed in a prone position. After sequential dilatations were performed under fluoroscopy, a 16.5 Fr or 21 Fr am Platz sheath was placed in the pelvicalyceal system. Ho: YAG Laser lithotripter (Sphinx, Lisa laser, USA) was used to fragment stones. According to the surgeon's decision, a JJ stent and/or a nephrostomy tube were placed at the final of the operation.

Primary outcome The primary outcome was the comparison of changes in haemoglobin and haematocrit values during two postoperative days with changes in intraoperative SpHb values and postoperative need for blood transfusion. SpHb was monitored throughout the surgery; however, the value of change before and immediately after surgery was a major concern. Blood samples were evaluated for Hb and Hct values on the first night and the second morning after surgery. Indications for blood transfusion were below 30% hematocrit level.

Secondary outcomes The effect on surgical outcomes was questioned by residual fragment (%) and postoperative complications. The effect on surgical practice was evaluated by operation time (minute) and visual score of the surgeon. At the end of the surgery, the assigned surgeon who was blind to the groups was asked to rate the visual clarity by a score pre-designed for arthroscopic surgeries as 'Bad-Medium, Good or Perfect'. A visual scoring from 1 to 10 was used, with 10 for the perfect image, 4-10 as good and 1-4 as bad-medium. We searched for bleeding, angioembolisation, infection, reoperation, and thrombotic complications, especially pulmonary emboli.

Statistical analysis and sample size calculation The mean sample size was calculated using the G Power 3.1 analysis program. The sample size was estimated at 90% power and 8% significance level, and it was determined that at least 20 patients per group were required to obtain a statistically significant value. Therefore, we included 25 patients in each group to prevent possible dropouts.

The Statistical Package for the Social Sciences version 27 (SPSS IBM Corp., Armonk, NY, USA) program was used. The normality of the distribution of the variables was checked by the Shapiro-Wilk test and Q-Q plots. The one-way ANOVA test or Kruskal-Wallis test was used for the comparison of continuous variables. Comparison between groups was performed with Tukey posthoc analysis. Qualitative data are shown as mean ± standard deviation or median (IQR). Quantitative data are shown as mean ± standard deviation values. The data were analyzed at a 95% confidence level.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old
* ASA I-III patients
* scheduled for PCNL surgery

Exclusion Criteria:

* tranexamic acid hypersensitivity
* history of subarachnoid haemorrhage
* previous cerebrovascular event
* a history of arterial-venous embolism or a tendency to thromboembolism
* abnormal liver function tests
* unstable cardiovascular disease
* acute or chronic renal failure
* the presence of any haematological disease and known colour blindness

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Hemoglobin decrease | postoperative 48 hours
  Hemoglobin decrease after postoperative first and second day relevant to preoperative values
Blood product requirement | postoperative 48 hours
  number of packed red blood cell use

SECONDARY OUTCOMES:
surgical visual score | intraoperative
  A visual scoring from 1 to 10 was used, with 10 for the perfect image, 4-10 as good and 1-4 as bad-medium

CONTACTS AND LOCATIONS:
Locations (1):
- Haseki Training and Research Hospital, Istanbul, Sultangazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ersin M, Demirel M, Buget MI, Edipoglu IS, Atalar AC, Ersen A. The effect of intravenous tranexamic acid on visual clarity during arthroscopic rotator cuff repair: A randomized, double-blinded, placebo-controlled pilot study. Acta Orthop Traumatol Turc. 2020 Nov;54(6):572-576. doi: 10.5152/j.aott.2020.19164. PMID 33423986
- [Result] Kim J, Alrumaih A, Donnelly C, Uy M, Hoogenes J, Matsumoto ED. The impact of tranexamic acid on perioperative outcomes in urological surgeries A systematic review and meta-analysis. Can Urol Assoc J. 2023 Jun;17(6):205-216. doi: 10.5489/cuaj.8254. PMID 36952300